CLINICAL TRIAL: NCT00171912
Title: Imatinib Mesylate in Patients With Various Types of Malignancies Involving Activated Tyrosine Kinase Enzymes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BAU12
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Hypereosinophilic Syndrome; Systemic Mastocytosis; Chronic Myelomonocytic Leukemia; Dermatofibrosarcoma
Keywords: Imatinib mesylate; tyrosine kinases; imatinib sensitivity; Diverse malignancies either associated with; or thought to be associated with; activated tyrosine kinase enzymes; including hypereosinophilic syndrome; systemic mastocytosis; chronic myelomonocytic leukaemia,; dermatofibrosarcoma protuberans and other diseases.; Not included:; patients with chronic myeloid leukemia,; some other types of leukemias (abl-mutated); some types of gastrointestinal stromal tumours (c-KIT-positive),; some systemic mastocytosis (if c-KIT D816V mutation),; brain,; prostate,; breast or lung cancers.
MeSH Terms: conditions — Hypereosinophilic Syndrome; Mastocytosis, Systemic; Leukemia, Myelomonocytic, Chronic; Dermatofibrosarcoma; Leukemia, Myelomonocytic, Juvenile; Lung Neoplasms | interventions — Imatinib Mesylate

ARMS (1):
- imatinib mesylate (STI571) (Experimental)
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate
  Other Names: STI571

SUMMARY:
This trial is for various types of malignancies which may depend on certain enzymes (tyrosine kinases) for growth. The objective of this study is to assess to what extent imatinib mesylate blocks these enzymes and to assess the effect on the malignancy.

DETAILED DESCRIPTION:
Condition

Diverse malignancies either associated with or thought to be associated with activated tyrosine kinase enzymes including hypereosinophilic syndrome systemic mastocytosis chronic myelomonocytic leukaemia, dermatofibrosarcoma protuberans and other diseases.

Not included:

Patients with chronic myeloid leukemia, some other types of leukemias (abl-mutated) some types of gastrointestinal stromal tumours (c-KIT-positive), some systemic mastocytosis (if c-KIT D816V mutation), brain, prostate, breast or lung cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Malignancy likely related to an activated tyrosine kinase enzyme sensitive to imatinib mesylate.
2. Spread of the disease to the rest of the body (confirmed by tissue sample) beyond the skin.
3. Malignant tissue showing activation of certain tyrosine kinases (ABL, ARG, KIT (CD117), or PDGF-R alpha or beta) & preferably within 6 weeks of entry.

Exclusion Criteria:

1. Certain leukaemias (abl-mutated), some gastrointestinal stromal tumours (c-KIT-positive) or certain systemic mastocytosis (if c- KIT D816V mutation).
2. A primary prostate, breast, lung or brain tumour,
3. Patient has previously been treated with imatinib mesylate except where treatment was more than 6 months previously and there is no suggestion of clinical resistance nor lack of response.

Other protocol-defined inclusion / exclusion criteria may apply.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy and the safety of imatinib mesylate therapy | 2 years

SECONDARY OUTCOMES:
To evaluate the effects of imatinib on quality of life and healthcare resource use | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, East Melbourne, Australia